CLINICAL TRIAL: NCT05484934
Title: Open Label Case Reports Investigating Wound Healing, Aesthetic Outcomes, and Patient Satisfaction Following Nipple-Areolar Complex (NAC) Reconstruction Using a Decellularized Donor NAC Graft (DCLNAC)
Brief Title: Investigate Wound Healing, Aesthetics & Pt Satisfaction Post NAC Reconstruction Using a Decellularized Donor NAC Graft
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: BioAesthetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BA002
Record Dates: First submitted 2022-07-13; First posted 2022-08-02 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Post-Mastectomy Breast Deformity (Disorder)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implant of acellular NAC graft (Experimental): The implantation of the NAC acellular graft for regenerative nipple areolar complex
  Interventions: Procedure: Regenerative post mastectomy surgery

INTERVENTIONS:
Procedure: Regenerative post mastectomy surgery — Implantation of the Nipple-Areolar Complex (NAC) Reconstruction Using a Decellularized Donor NAC Graft (DCLNAC)
  Other Names: Implantation of the NAC graft

SUMMARY:
To evaluate the wound healing response following nipple-areolar complex (NAC) reconstruction with a decellularized donor NAC graft (DCLNAC)

DETAILED DESCRIPTION:
Primary Objective

• To evaluate the wound healing response following nipple-areolar complex (NAC) reconstruction with a decellularized donor NAC graft (DCLNAC).

Secondary Objectives

* To evaluate nipple dimensions and vascularization up to 12 months following nipple reconstruction using DCLNAC.
* To evaluate patient satisfaction and well-being up to 12 months following nipple reconstruction using DCLNAC.

Exploratory Objectives

* To assess operative time and physician preference for either the DCLNAC or the standard of care (SOC) surgical NAC reconstruction procedures.
* To evaluate nipple sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* General Criteria:

  * Females age >18 and <65 years old. Women of childbearing potential must agree to use an acceptable method of contraception for one month prior to DCLNAC implantation, and until the graft is 100% healed. Acceptable forms of birth control include abstinence, birth control pills, or any double combination of: intrauterine device (IUD), male or female condom, diaphragm, sponge, and cervical cap. Nonchildbearing potential for women is defined as postmenopausal (last natural menses greater than 12 months) or undergone a documented bilateral tubal ligation or hysterectomy. If last natural menses less than 12 months, a serum FSH value confirming post-menopausal status can be employed.
  * Patient agrees to sleep on back until study tissue products are healed
  * Patient agrees to abstain from aspirin, alcohol, or excessive caffeine until study tissue products are healed
  * Patient agrees to not undergo NAC tattooing until completing study
  * Patient can understand and willing to sign informed consent
  * Patient desires bilateral nipple reconstruction with DCLNAC
  * Subjects must be capable of providing written informed consent to the study procedures and for use of protected health information [Health Insurance Portability and Accountability Act (HIPAA), if applicable]

    * Specific Criteria

Group A:

* Patient had a bilateral mastectomy with no radiation therapy
* Patient has undergone a bilateral autologous breast reconstruction a minimum of 3 months prior to enrolling in the study

Group B:

* Patient had a unilateral mastectomy with no radiation therapy
* Patient has undergone a unilateral autologous breast reconstruction a minimum of 3 months prior to enrolling in the study

Group C:

* Patient had a bilateral mastectomy and received radiation unilaterally
* Patient has undergone a bilateral autologous breast reconstruction a minimum of 3 months prior to enrolling in the study

Group D:

- Patient had unilateral or bilateral mastopexy (with or without augmentation) or reduction mammaplasty and suffered nipple complications (i.e., necrosis, projection loss)

Group E:

* Patient had unilateral or bilateral mastectomy
* Patient had unilateral or bilateral autologous breast reconstruction a minimum of 3 months prior to enrolling in the study
* Patient did not receive radiation to the autologously reconstructed breast
* Patient had unilateral or bilateral nipple reconstruction that failed (i.e., necrosis, projection loss)

Group F:

- Implant based reconstruction

Exclusion Criteria:

* Patient has a history of delayed wound healing
* Patient has a history of Vitamin C deficiency
* BMI<18.5 or >40 kg/m2
* Patient has a history of allergic reaction to any decellularized biologic matrix product
* Patient is currently smoking or using tobacco or nicotine products (i.e., patch, gum, vaping or nasal spray) or has used such products in the past 6 months
* Patient is currently receiving bilateral breast radiation or completed less than 3 months prior to screening
* Patient has any systemic disease that would impede wound healing, such as diabetes or connective tissue disorders
* Patient is pregnant, breastfeeding or planning to become pregnant during the study period
* Patient has any type of disease or disorder that in the investigator's opinion would make the patient unfit for the study, including active infection anywhere in the body.
* Acute mastitis in either breast
* History of an autoimmune disorder
* Use of any medications currently or in the past 3 months that would impair wound healing, such as long-term use of systemic steroids (inhaled, limited topical, short-term oral use and intra-articular steroids are acceptable)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 36 (Estimated)
Dates: Start 2022-09-21 (Actual); Primary Completion 2024-08-07 (Estimated); Study Completion 2024-10-07 (Estimated)

PRIMARY OUTCOMES:
Time to complete healing (graft >99% re-epithelialized) | 3 months
  To evaluate the time to complete healing following NAC reconstruction with DCLNAC.
Healing of the nipple (VAS=Visual Analog Scale) epithelialization | 3 months
  epithelialization (0-100% VAS)
Healing of the nipple (VAS=Visual Analog Scale) granulation | 3 months
  granulation (0-100% VAS)
Healing of the nipple (VAS=Visual Analog Scale) ischemia/necrosis | 3 months
  ischemia/necrosis (0-100% VAS)
Healing of the nipple (VAS=Visual Analog Scale) dehiscence | 3 months
  dehiscence (0-100% VAS)
Healing of the nipple (VAS=Visual Analog Scale) overall healing | 3 months
  overall healing (0-100% VAS)
Healing of the nipple (infection) A. no infection B. hyperemia (no infection) C. cellulitis (superficial infection D. abscess or purulent infection | 3 months
  As above

SECONDARY OUTCOMES:
Nipple projection | 12 months
  Distance from breast mound to tip in millimeters using depth gauge.
Vascularization by presence of bleeding | 12 months
  vascularization by presence of bleeding using a lancet device
Evaluate patient satisfaction and well-being preoperatively and serially | 12 months
  Use of a standardized postoperative survey with a LIKERT (numerical) scale up to 12 months following reconstruction.

OTHER OUTCOMES:
Operative time in minutes | 12 months
  One hour
Physician Preference and Impressions | 12 months
  Using a standardized survey (0-10 VAS Scale)
Nipple sensitivity up to 12 months | 12 months
  Using Semmes Weinstein Monofilament

CONTACTS AND LOCATIONS:
Overall Officials: Roger Morgan, MD, Study Chair — MedSurgPI, LLC
Locations (1):
- St. Charles Surgical Hospital, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No